CLINICAL TRIAL: NCT06659159
Title: Effects of Beginning a GLP1-Agonist Therapy on Residual Gastric Content and Gastric Emptying: a Prospective Ultrasound Approach with Focus on Perioperative Aspiration Risk.
Brief Title: Effects of Beginning a GLP1-Agonist Therapy on Residual Gastric Content and Gastric Emptying
Acronym: GLP-1
Status: Not yet recruiting | Type: Observational
Sponsor: Sascha Battig (Other)
Responsible Party: Sponsor-Investigator, Sascha Battig, Prof. Dr. med. Michael Ganter, Klinik Hirslanden, Zurich
Organization: Klinik Hirslanden, Zurich (Other)
Other Study IDs: Effects of beginning a GLP1; Hirslanden Klinik (Other Grant/Funding Number: Hirslanden Klinik, Zurich)
Record Dates: First submitted 2024-10-04; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Aspiration During Anaesthetic Induction
Keywords: Pulmonary aspiration; Gastric ultrasound; GLP-1; Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GLP-1, New Therapy: Indication, prescription and dosage is determined independently of the study by the endocrinologist/obesity specialist, who is also part of the study team. Since the first gastric ultrasound will take place directly before the initiation of the GLP-1 Agonist therapy, the patients will serve as their own control group/baseline.
  Interventions: Diagnostic Test: Gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — The sequence in which the study is conducted will be as follows, the first examination (baseline examination) will take place immediately before the appointment and prescription of GLP-1 Analoga (before the first injection). During the examination the gastric content (quality/quantity) will be determined, secondly, a baseline for gastric emptying time after oral intake of 500ml of water is collected (patient drinks water, the stomach emptying will simultaneously be tracked with gastric ultrasound).
  In accordance with the first endocrinological control examination (6-8 weeks after therapy initiation) the same gastric ultrasound examination is performed.

SUMMARY:
This project explores the elevated risk of pulmonary aspiration during anesthesia in patients undergoing GLP-1 agonist therapy, which prolongs gastric emptying. Despite standard fasting guidelines (6 hours for solids, 2 hours for liquids), some patients still experience aspiration, indicating that GLP-1 therapy may heighten risk. The American Society of Anesthesiologists has advised pausing GLP-1 therapy before surgery, but this recommendation has faced criticism for being too broad. More data on this issue is needed, particularly concerning the effect of tachyphylaxis (reduced drug response over time) on gastric emptying.

The study proposes using gastric ultrasound as a non-invasive tool to evaluate residual gastric content and categorize patients by their aspiration risk. The study will assess the stomach's content and gastric emptying time in patients both before and after starting GLP-1 therapy, comparing results under standard fasting conditions.

The project is a national, single-center, prospective observational study targeting 50 patients, examining factors like patient demographics, GLP-1 therapy details, and gastrointestinal side effects. Data collection will occur through baseline and follow-up sonographic exams before and after therapy initiation. The study aims to improve perioperative management strategies by clarifying the risks associated with GLP-1 therapy

DETAILED DESCRIPTION:
This project investigates the risk of pulmonary aspiration during anesthesia in patients undergoing treatment with GLP-1 agonists, a class of medications that prolong gastric emptying and are commonly used for obesity and diabetes management. Pulmonary aspiration remains a significant cause of morbidity and mortality in anesthesia-related complications, and patients with delayed gastric emptying are at higher risk. Recent reports suggest that patients taking GLP-1 agonists may be at increased risk for aspiration, even when adhering to standard perioperative fasting guidelines (6 hours for solids, 2 hours for liquids).

The American Society of Anesthesiologists (ASA) has issued a warning about the potential risk of aspiration in patients on GLP-1 agonist therapy, recommending pausing the medication before surgery. However, this recommendation has been criticized for being too broad, given the lack of comprehensive data on the exact impact of GLP-1 agonists on gastric emptying and aspiration risk. Since many patients treated with GLP-1 agonists are already at higher risk of aspiration due to comorbidities like obesity and diabetes, understanding how this therapy further affects gastric function is crucial. There are also indications of a "tachyphylaxis" effect, where patients develop tolerance to the drug's impact over time, but its effect on gastric emptying and perioperative aspiration risk is not well understood.

Study Rationale and Objectives

The primary aim of this study is to assess whether patients undergoing GLP-1 agonist therapy have a higher likelihood of a full stomach after the recommended fasting intervals. Additionally, the study aims to evaluate the time taken for gastric emptying in these patients, focusing on the clearance of 500 ml of water.

Study Design

The project is a national, single-center, prospective observational study that will include approximately 50 patients who are starting GLP-1 agonist therapy. Patients will serve as their own control group by undergoing gastric ultrasound before beginning treatment and then again 6-8 weeks after therapy initiation. If therapy is continued, a follow-up ultrasound will occur around 5 months later.

The ultrasound examinations will measure both the gastric content (solid, liquid, or empty) and the cross-sectional area (CSA) of the gastric antrum to estimate gastric volume. These measurements will provide insight into whether patients on GLP-1 agonists have prolonged gastric emptying, contributing to the risk of aspiration during surgery.

Study Population and Procedures

The study population will consist of patients prescribed GLP-1 agonists for obesity, diabetes, or lifestyle reasons. Inclusion criteria include adults beginning a new GLP-1 therapy regimen, while exclusion criteria rule out patients with known gastrointestinal disorders, previous GI surgery, pregnancy, and those at high risk for hypoglycemia due to other medications like sulfonylureas or insulin.

Recruitment will occur through collaboration with the Adipositas und StoffwechselZentrum Hirslanden Zurich, where GLP-1 agonists are regularly prescribed. Patients will be contacted by phone to provide initial study information, and written informed consent will be obtained before the baseline examination. A demographic and medical history will also be collected at the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Beginning a new treatment with GLP-1 Agonists. Indication and prescription determined by an endocrinologist/obesity specialist
* Signed informed consent

Exclusion Criteria:

* Known pregnancy, known lactation
* Underage (< 18 years)
* Absence of informed consent (missing or inability to provide)
* Anomalies of the gastrointestinal tract
* Known illnesses of the gastrointestinal tract
* Previous surgery of the gastrointestinal tract
* Elevated risk for hypoglycaemia (Sulfonylurea or Insulin)
* No investigator with completed structural education in gastric sonography is available
* Lack of intention to respect the fasting intervals and predefined standardised meals for the sonographic examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GLP-1 Therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric content | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Sonographic assessment of the gastric content (quality and quantity) after a standardised meal and regular perioperative fasting interval (at least 6 hours for solids and 2 hours for liquids) before initiation and once 6-8 weeks after GLP-1 therapy initiation

SECONDARY OUTCOMES:
Gastric emptying time | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Sonographic measurement of gastric emptying time for 500ml of water before and during GLP-1 therapy. Gastric emptying time is measured with a continuous ultrasound examination. The variable of interest is once again the CSA of the gastric antrum and the time until the baseline from before water consumption is reached once again.
Number of empty stomachs | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Absolute number of empty stomachs after adhering to standardised perioperative fasting intervals (6 hours for solids and 2 hours for liquids) before and once (if therapy is continued: twice) during GLP-1 Agonist therapy
BMI | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Demographic data of the patient: BMI
Gallbladder stones | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Presence of gallbladder stones (cholecystolithiasis)
Co-morbidities | At the baseline examination at the first endocrinologic appointment
  Demographic data of the patients: Comorbidities
Side effects GLP-1 | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Collection of all side-effects of the GLP-1 therapy
Discontinuation GLP-1 | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  Number and reason for discontiuation of GLP-1 therapy
Co-medication | baseline examination at the first endocrinologic appointment the second examination/data collection will be at the regular endocrinologic control examination 6-8 weeks after therapy initiation. Final examination is 5 months after therapy start
  For gastric emptying relevant co-medications

IPD SHARING:
Plan to Share IPD: No